CLINICAL TRIAL: NCT04056026
Title: A Single Dose FMT Infusion From a Healthy Family Donor Via Colonoscopy as an Adjunct to Keytruda for the Benefit of Improving Efficacy of Immunotherapy for Metastatic Mesothelioma
Brief Title: A Single Dose FMT Infusion as an Adjunct to Keytruda for Metastatic Mesothelioma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: ProgenaBiome (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ProgenaBiome-001
Record Dates: First submitted 2019-08-07; First posted 2019-08-14 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fecal Microbiota Transplant (Experimental): The patient will undergo fecal microbiota transplant. The 600cc of donor stool will be transplanted by colonoscopy.
  Interventions: Biological: Fecal Microbiota Transplant

INTERVENTIONS:
Biological: Fecal Microbiota Transplant — Fecal material from a healthy family donor will be transplanted into the patient via colonoscopy
  Other Names: FMT

SUMMARY:
The investigators propose to ensure a favorable gut microbiome by fecal microbiota transplant to enhance the efficacy Keytruda

DETAILED DESCRIPTION:
Studies have shown that a favorable microbiome can be the difference between response and non-response of certain cancer treatments such as PD-1 blockade inhibitors. As such the investigators propose to ensure a favorable microbiome in this patient by fecal microbiota transplant to enhance the efficacy of such a drug, Keytruda.

ELIGIBILITY:
Inclusion Criteria:

* Patient with metastatic mesothelioma deemed a candidate for PD-1 blockade inhibitor therapy

Exclusion Criteria:

* Patient unable/unwilling to comply with protocol
* Patient deemed not a candidate for PD-1 Blockade inhibitor therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Five years
  The time from transplant that the patient's tumors remain stable or shrink.

CONTACTS AND LOCATIONS:
Locations (1):
- ProgenaBiome, Ventura, California, United States